CLINICAL TRIAL: NCT01615601
Title: PREZISTA or INTELENCE Switch Evaluation in Virologically Suppressed Patients Naïve to Darunavir or Etravirine and Who Are Intolerant of Their Current or Prior Combination Antiretroviral Therapy Regimen: A Phase IV, Open-label, Multicentre Observational Trial
Brief Title: An Observational Study to Evaluate Tolerability of PREZISTA or INTELENCE in HIV-1 Infected Patients
Acronym: POISE
Status: Completed | Type: Observational
Sponsor: Janssen Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR018595; TMC114HIV4068 (Other: Janssen Inc.)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: Human Immunodeficiency Virus; HIV; HIV-1; HIV type 1; Darunavir; PREZISTA; Etravirine; INTELENCE; HIV symptom Distress Module; HIV-SDM; Antiretroviral therapy; HIV Symptom Index (HSI),
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir; etravirine; Ritonavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- darunavir (PREZISTA): PREZISTA co-administered with 100 mg ritonavir as per Canadian Product Monograph. (Observational Study)
  Interventions: Drug: darunavir (PREZISTA); Drug: ritonavir
- etravirine (INTELENCE): INTELENCE co-administered with other antiretroviral medicinal products as per Canadian Product Monograph (Observational Study)
  Interventions: Drug: etravirine (INTELENCE); Drug: Other antiretroviral medications

INTERVENTIONS:
Drug: darunavir (PREZISTA) — Form = tablet, route = oral, Units = mg, number = 800 administered once daily
  Groups: darunavir (PREZISTA)
Drug: etravirine (INTELENCE) — Form = tablet, route = oral, Unit = mg, number = 200, administered twice daily
  Groups: etravirine (INTELENCE)
Drug: ritonavir — Form = tablet/capsule, route = oral, Units = mg, number = 100 administered once daily
  Groups: darunavir (PREZISTA)
Drug: Other antiretroviral medications — Given as per Canadian Product Monograph
  Groups: etravirine (INTELENCE)

SUMMARY:
The purpose of this study is to evaluate tolerability of darunavir (PREZISTA) or etravirine (INTELENCE) in patients infected with human immunodeficiency virus type 1 (HIV-1) who are naïve to these medications and in patients who have experienced tolerability issues on their current or prior combination antiretroviral therapy (cART). The tolerability is evaluated by switching the patients from their previous or current combination antiretroviral therapy (cART) to either darunavir or etravirine.

DETAILED DESCRIPTION:
This is an open label (all people know the identity of the intervention.), multicenter (study conducted at multiple sites), observational study (individuals are observed for certain outcomes) of darunavir and etravirine in patients infected with HIV-1 who are naïve to these medications and who have experienced tolerability issues on their current or prior combination antiretroviral therapy (medicines used for treatment of HIV). PREZISTA is indicated for naïve HIV patients (someone who has never used HIV drugs) and treatment-experienced HIV patients and INTELENCE is indicated for treatment-experienced patients who have failed prior therapy and have HIV-1 strains resistant to multiple antiretroviral agents (HIV-1 strains are able to survive the exposure of the multiple antiretroviral agents), including Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTIs). In this study patients will receive either darunavir (PREZISTA) or etravirine (INTELENCE) and physician selected optimized background agents (other antiretroviral medicines), as permitted by the local formulary and supported by the current Canadian Product Monograph. 90 patients will participate in this study (75 Patients planned for the darunavir group and 15 patients planned for the etravirine group). The total duration of the study will be 24 weeks. Safety and tolerability will be evaluated at screening (14 days prior to Day 1), baseline (patient's medical status before any treatment or research is done) at Day 1, Week 4, Week 12 and Week 24. Tolerability will be evaluated using HIV Symptom Distress Module (HIV-SDM) also referred to as the HIV Symptom Index (HSI) which is a self-completed questionnaire to evaluate symptoms and measure the presence and bothersomeness of side effects commonly seen with HIV and antiretroviral treatment over the last 4 weeks (20 questions about all symptoms which the patient might have had during the past four weeks). Higher scores indicate the presence of more symptoms and/or a greater degree of distress related to the 20 symptoms. In HIV-SDM data is collected to see the benefit of switching to either darunavir or etravirine.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented HIV-1 infection
* Have 1 or more significant symptoms with at least grade 2 toxicity on the Division of AIDS Toxicity "DAIDS grading scale" on current or prior combination antiretroviral therapy (cART) regimen (current or prior cART including regimens consisting of 2 Nucleoside reverse transcriptase inhibitors (NRTIs) and a third agent with the exception of darunavir or etravirine)
* Have stable response to current cART ie, have an HIV-plasma viral load [number of virus in blood] at screening <400 copies/mL (undetectable) or last plasma viral load on prior regimen within the previous 6 months <400 copies/mL)
* Must not have resistance to Primary HIV protease inhibitor medicines

Exclusion Criteria:

* Has been Infected with HIV-2 - Has received previous treatment with darunavir or etravirine or non-HAART (Highly Active Antiretroviral Therapy) regimen
* Has had prior virologic failure to 2 or more regimens or single virologic failure on prior cART
* Has a documented resistance to darunavir and etravirine
* Is currently using any drug contraindicated in the current Canadian Product Monograph for darunavir or etravirine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients infected with human immunodeficiency virus type 1 who have experienced tolerability issues on their current or prior ccombination antiretroviral therapy regimen and for whom a regimen including darunavir and/or etravirine is clinically indicated.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the patient's total score of the HIV Symptom Distress Module (HIV-SDM) | Baseline (Day 1), Week 4, 12 and 24
  HIV-SDM is a questionnaire consisting of 20 questions related to all the symptoms which the patient might have had during the past four weeks. For each question patient has to select appropriate answer related to the symptoms: "0 = I do not have this symptom; 1 = I have this symptom and it doesn't bother me; 2 = it bothers me a little; 3 = it bothers me; 4 = it bothers me a lot". Total score of HIV-SDM is then calculated for all the 20 items.

SECONDARY OUTCOMES:
Number of participants with Maintenance/achievement of virologic suppression at Week 24 | Baseline and Week 24
  Virologic suppression is decrease in the number of virus in blood. Number of participants with virologic suppression (who achieved virologic suppression) as well as the Number of participants who maintained virologic suppression will be summarized.
Number of participants with disappearance by Week 4 of at least one bothersome symptom identified at baseline by patient on HIV-SDM | Baseline and Week 4
  The bothersome symptoms (defined as those reported as 'It bothers me a lot' or 'It bothers me') at baseline will be identified for each patient. The number of participants who report the disappearance of at least one of the bothersome symptoms (eg, reported as 'It bothers me a little', 'It does not bothers me', 'I do not have the symptom') by Week 4 will be summarized.
Number of participants with maintenance of disappearance by Week 12 and Week 24 of at least one bothersome symptom identified at baseline by patient on HIV-SDM | Baseline, Week 12 and Week 24
  The number of participants who report the maintenance of the disappearance of at least one of the bothersome symptoms (eg, reported as It bothers me a little, 'It does not bothers me', 'I do not have the symptom') at Week 12 and Week 24 will be summarized.
Number of participants with Maintenance/increase in CD4 cell count. | Baseline and Week 24
  CD4 cells (a type of white blood cells) are circulating in blood and gives an idea of how strong the HIV positive person's immune system really is. The values of CD4 cell counts will be summarized using mean, standard deviations, minimum and maximum at baseline and Week 24. In addition, the number of participants with maintenance or increase in CD4 cell counts will be summarized.
Comparison of change in HIV-SDM scores between those participants who were on or off ARTs at baseline | Baseline, Week 4, Week 12 and Week 24
  On and off ARTs is patients taking HIV medications and patients not taking HIV medications. The HIV-SDM change from baseline scores will be summarized using basic statistics (mean, standard deviations, minimum and maximum) by whether the patient is on or off ART at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Inc. Clinical Trial, Study Director — Janssen Inc.
Locations (1):
- Vancouver, Canada